CLINICAL TRIAL: NCT00353470
Title: Dynamic Treatment vs. CBT for Panic Disorder
Brief Title: Comparison of Psychotherapy Programs to Treat Panic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH070918 (NIH); R01MH070664 (NIH)
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Anxiety Disorders; Panic Disorder; Agoraphobia
Keywords: PD; CBT; PFPP
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Agoraphobia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive panic focused psychodynamic psychotherapy for 12 weeks
  Interventions: Behavioral: Panic focused psychodynamic psychotherapy (PFPP)
- 2 (Active Comparator): Participants will receive cognitive behavioral therapy-panic control treatment for 12 weeks
  Interventions: Behavioral: Cognitive behavioral therapy
- 3 (Active Comparator): Participants will receive applied relaxation training for 12 weeks
  Interventions: Behavioral: Applied relaxation training (ART)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT for panic disorder will include 19 to 24 sessions over 12 weeks.
  Other Names: Panic control treatment
  Arms: 2
Behavioral: Applied relaxation training (ART) — ART with exposure protocol will include 19 to 24 sessions over 12 weeks.
  Other Names: ART
  Arms: 3
Behavioral: Panic focused psychodynamic psychotherapy (PFPP) — PFPP will include 19 to 24 sessions over 12 weeks.
  Arms: 1

SUMMARY:
This study will determine the relative effectiveness of three psychotherapies in treating people with a panic disorder.

DETAILED DESCRIPTION:
Panic disorder (PD) is a debilitating anxiety disorder. It is characterized by unexpected and repeated episodes of intense fear, accompanied by serious physical symptoms, such as chest pain, heart palpitations, shortness of breath, dizziness, or abdominal stress. Available treatments for PD include medication therapy and cognitive behavioral therapy (CBT), a type of psychotherapy that teaches people how to view panic attacks differently and how to reduce anxiety. Approximately 30% of patients refuse medication, however, and nearly 50% do not achieve remission with CBT alone. Therefore, there is a pressing need for additional non-pharmacologic treatment methods. Panic-focused psychodynamic psychotherapy (PFPP) and applied relaxation training (ART) are among some of the other available treatments for PD. During ART, individuals are taught to relax their muscles while being exposed to increasingly frightening situations. PFPP combines elements of CBT with other, more extensive approaches aimed at determining the anxiety's origin and at finding ways to reduce it. This study will compare the effectiveness of PFPP, CBT, and ART in treating PD.

Participants in this single blind study will be randomly assigned to receive PFPP, CBT, or ART for 12 weeks. All participants will attend between 19 and 24 treatment sessions over the course of the study. Upon completing the study, participants will attend monthly follow-up visits for an additional 12 months. Participants assigned to ART who have not responded by the end of treatment may opt to receive PFPP or CBT. Outcomes will be assessed using a variety of scales to determine depression and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for primary PD with or without agoraphobia
* History of at least one spontaneous panic attack per week within the month prior to study entry

Exclusion Criteria:

* Active substance dependence within 6 months prior to study entry
* Lifetime history of any psychotic disorder, including bipolar disorder
* Acutely suicidal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-09; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Milrod, MD, Principal Investigator — Weill Medical College of Cornell University; Jacques P. Barber, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, New York, New York
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Milrod B, Leon AC, Busch F, Rudden M, Schwalberg M, Clarkin J, Aronson A, Singer M, Turchin W, Klass ET, Graf E, Teres JJ, Shear MK. A randomized controlled clinical trial of psychoanalytic psychotherapy for panic disorder. Am J Psychiatry. 2007 Feb;164(2):265-72. doi: 10.1176/ajp.2007.164.2.265. PMID 17267789
- [Background] Milrod BL, Leon AC, Barber JP, Markowitz JC, Graf E. Do comorbid personality disorders moderate panic-focused psychotherapy? An exploratory examination of the American Psychiatric Association practice guideline. J Clin Psychiatry. 2007 Jun;68(6):885-91. doi: 10.4088/jcp.v68n0610. PMID 17592913
- [Result] Milrod B, Chambless DL, Gallop R, Busch FN, Schwalberg M, McCarthy KS, Gross C, Sharpless BA, Leon AC, Barber JP. Psychotherapies for Panic Disorder: A Tale of Two Sites. J Clin Psychiatry. 2016 Jul;77(7):927-35. doi: 10.4088/JCP.14m09507. PMID 27464313
- [Derived] Keefe JR, Chambless DL, Barber JP, Milrod BL. Predictors and moderators of treatment dropout in cognitive-behavioral and psychodynamic therapies for panic disorder. Psychother Res. 2021 Apr;31(4):432-442. doi: 10.1080/10503307.2020.1784487. Epub 2020 Jun 25. PMID 32584211
- [Derived] Barber JP, Milrod B, Gallop R, Solomonov N, Rudden MG, McCarthy KS, Chambless DL. Processes of therapeutic change: Results from the Cornell-Penn Study of Psychotherapies for Panic Disorder. J Couns Psychol. 2020 Mar;67(2):222-231. doi: 10.1037/cou0000417. PMID 32105128
- [Derived] Keefe JR, Huque ZM, DeRubeis RJ, Barber JP, Milrod BL, Chambless DL. In-session emotional expression predicts symptomatic and panic-specific reflective functioning improvements in panic-focused psychodynamic psychotherapy. Psychotherapy (Chic). 2019 Dec;56(4):514-525. doi: 10.1037/pst0000215. Epub 2019 Mar 14. PMID 30869969
- [Derived] Solomonov N, Falkenstrom F, Gorman BS, McCarthy KS, Milrod B, Rudden MG, Chambless DL, Barber JP. Differential effects of alliance and techniques on Panic-Specific Reflective Function and misinterpretation of bodily sensations in two treatments for panic. Psychother Res. 2020 Jan;30(1):97-111. doi: 10.1080/10503307.2019.1585591. Epub 2019 Mar 1. PMID 30821630
- [Derived] Suarez-Jimenez B, Zhu X, Lazarov A, Mann JJ, Schneier F, Gerber A, Barber JP, Chambless DL, Neria Y, Milrod B, Markowitz JC. Anterior hippocampal volume predicts affect-focused psychotherapy outcome. Psychol Med. 2020 Feb;50(3):396-402. doi: 10.1017/S0033291719000187. Epub 2019 Feb 18. PMID 30773148
- [Derived] McCarthy KS, Chambless DL, Solomonov N, Milrod B, Barber JP. Twelve-Month Outcomes Following Successful Panic-Focused Psychodynamic Psychotherapy, Cognitive-Behavioral Therapy, or Applied Relaxation Training for Panic Disorder. J Clin Psychiatry. 2018 Sep 11;79(5):17m11807. doi: 10.4088/JCP.17m11807. PMID 30256548
- [Derived] Solomonov N, McCarthy KS, Gorman BS, Barber JP. The Multitheoretical List of Therapeutic Interventions - 30 items (MULTI-30). Psychother Res. 2019 Jul;29(5):565-580. doi: 10.1080/10503307.2017.1422216. Epub 2018 Jan 16. PMID 29336228

RESULTS

PARTICIPANT FLOW:
Groups:
- PFPP: Participants will receive panic focused psychodynamic psychotherapy for 12 weeks
  Panic focused psychodynamic psychotherapy (PFPP): PFPP will include 19 to 24 sessions over 12 weeks.
- C.B.T.: Participants will receive cognitive behavioral therapy-panic control treatment for 12 weeks
  Cognitive behavioral therapy: CBT for panic disorder will include 19 to 24 sessions over 12 weeks.
- A.R.T.: Participants will receive applied relaxation training for 12 weeks
  Applied relaxation training (ART): ART with exposure protocol will include 19 to 24 sessions over 12 weeks.
Period: Overall Study
Arm/Group | PFPP | C.B.T. | A.R.T.
Started | 81 | 81 | 39
Completed | 61 | 61 | 23
Not Completed | 20 | 20 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PFPP | C.B.T. | A.R.T. | Total
Number analyzed (Participants) | 81 | 81 | 39 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 81 | 39 | 201
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.2) | 39.3 (12.9) | 36 (12) | 38.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 46 | 32 | 136
  Male | 23 | 35 | 7 | 65
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 39 | 201

OUTCOME MEASURES:

1. Primary Outcome: Panic Disorder Severity Scale
Description: A composite score of panic severity. High value = 28, lowest value =0. Higher=worse
Time Frame: 12 weeks
Population: one subject was eliminated from analyses with DSMB consent as they lied about symptoms at intake and did not meet inclusion criteria
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 80 | 81 | 39
score on a scale | 6.72 (4.49) | 5.78 (3.48) | 7 (2.94)
Statistical Analysis 1: Comparison: PFPP vs C.B.T. vs A.R.T; Power: to detect a between-group effect size of 0.45, for statistical power of 0.80, 56 patients for PFPP or CBT vs. 28 for ART were required. Response rates at termination were calculated by chi-square in the full ITT sample using LOCF; Test type: Superiority; p > 0.16, Chi-squared; shared parameters model = -.56, Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: PFPP vs C.B.T. vs A.R.T; Test type: Superiority; p < .05, Mixed Models Analysis

2. Secondary Outcome: Sheehan Disability Scale
Description: Level of psychosocial functional impairment. highest value=30, lowest value =0, higher numbers indicate greater dysfunction
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 78 | 79 | 38
score on a scale | 6.4 (6.74) | 6.28 (5.89) | 6.9 (4.43)

3. Secondary Outcome: Clinical Global Impressions Scale
Description: Clinical assessment of severity of impairment. Minimum value=1, maximum value =6; high scores worse
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 79 | 77 | 38
units on a scale | 2.17 (1.28) | 2.16 (0.90) | 2.38 (0.92)

4. Secondary Outcome: Hamilton Depression Rating Scale
Description: Level of state depression. scale 0-81, 0 symptom free, 81 worst severity
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 79 | 81 | 39
units on a scale | 11.37 [0 to 81] | 10.18 [0 to 81] | 11.55 [0 to 81]

5. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: level of state anxiety. 0=symptom free, 56 most severe
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 79 | 81 | 39
units on a scale | 7.97 (6.13) | 7.87 (5.89) | 6.30 (3.2)

6. Secondary Outcome: Anxiety Disorder Sensitivity Index
Description: Anxiety disorder sensitivity index measures Sensitivity to physical symptoms of anxiety (scores range from 0-64). 0= no anxiety, 64 =maximum anxiety
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 79 | 77 | 38
score on a scale | 27.07 (12.77) | 17.71 (9.87) | 19.09 (12.28)

7. Secondary Outcome: Brief Body Sensitivity Interpretation Questionnaire (BBSIQ)
Description: The BBSIQ measures how physically sensitive the person is to physical symptoms of anxiety; (scores range 0-63) 0= no anxiety; 63= highest levels of physical anxiety
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 73 | 79 | 37
score on a scale | 1.80 (0.39) | 1.62 (0.31) | 1.70 (0.27)

8. Secondary Outcome: Panic-Specific Reflective Function
Description: Ability to reflect on the emotional meaning of panic symptoms. scored -1 to 9, high numbers better
Time Frame: 12 weeks
Population: Data is presented for those subjects from whom data was collected for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFPP | C.B.T. | A.R.T.
Number analyzed (Participants) | 79 | 78 | 38
units on a scale | 4.67 (1.11) | 3.67 (1.15) | 3.20 (1.03)

ADVERSE EVENTS:
Time Frame: Subjects assessed for AEs for three months of therapy, 3 months of crossover (if eligible) and 12 months of follow-up; 15-18 months
Arm/Group | PFPP | C.B.T. | A.R.T.
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81 | 2/39
Other Adverse Events (participants affected / at risk) | 0/81 | 0/81 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PFPP (N=81) | C.B.T. (N=81) | A.R.T. (N=39)
hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 2/2 (2) — Psychiatric hospitalization required-1 pt with PTSD and depression; 1 pt developed psychotic depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No